CLINICAL TRIAL: NCT04236076
Title: Assessing Exercise Capacity After PulseHaler™ Treatment in Chronic Obstructive Lung Disease (GOLD) II-IV of Chronic Obstructive Pulmonary Disease (COPD) Patients
Brief Title: Assessing Exercise Capacity After PulseHaler™ Treatment in GOLD II-IV COPD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Respinova LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PH-03
Record Dates: First submitted 2019-12-18; First posted 2020-01-22 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2019-12

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PulseHaler™ (Experimental): Patients will receive PulseHaler for home treatment
  Interventions: Device: PulseHaler
- Sham PulseHaler - CONTROL group (Sham Comparator): Patients will receive Sham device for home treatment
  Interventions: Device: Sham - control

INTERVENTIONS:
Device: PulseHaler — PulseHaler™ is a pulsating positive expiratory pressure ventilation device for treatment of COPD. PulseHaler™ is pre-programmed to deliver airflow at pre-defined frequencies, ranging from 3.5 Hertz (Hz) to 55Hz, and for pre-defined lengths of time.
  Arms: PulseHaler™
Device: Sham - control — Sham device has the same look as PulseHaler and is set to deliver nominal pressure but it does not contain the active pulsating components.
  Arms: Sham PulseHaler - CONTROL group

SUMMARY:
Prospective, sham controlled, interventional study to evaluate the extent to which PulseHaler improves the functional status of Chronic Obstructive Lung Disease (GOLD) II-IV Chronic obstructive pulmonary disease (COPD) patients.

DETAILED DESCRIPTION:
PulseHaler™ is a pulsating positive expiratory pressure ventilation device for treatment of COPD . PulseHaler™ is pre-programmed to deliver airflow at pre-defined frequencies and for pre-defined lengths of time.

The study is intended to evaluate the extent to which PulseHaler improves the functional status of GOLD II-IV COPD patients after 4 weeks of treatment 3x / day.

And To evaluate the extent to which improvements are maintained over a subsequent 2 weeks when treatments are tapered to 1x daily.

ELIGIBILITY:
Inclusion Criteria:

* Investigator confirmation of GOLD II-IV COPD
* Successful completion of Incremental Exercise Test (IET)
* FEV1 < 60% predicted
* Post-bronchodilator FEV1/FVC ≤ 0.7
* 55-75 years old
* Signed informed consent by subject (required cognitive capacity)

Exclusion Criteria:

* SpO2<80% at IET
* Unable to achieve a CWR test duration at visit 2 between 3 and 8 minutes
* Exercise limitation unrelated to diagnosis of COPD
* Systemic (oral, IV, IM) steroid use for acute exacerbation in the 30 days prior to screening
* Baseline CAT Score <10
* Women at the age of fertility, who are pregnant, or plan pregnancy, or do not use contraceptives
* Severe cardiac disease, e.g., Congestive Heart Failure grade , hemodynamic instability,
* Acute myocardial infarction within last 3 months
* Coronary artery bypass graft within last 3 months
* Epilepsy, raised intracranial pressure, acute sinusitis or nosebleed
* Pulmonary embolism, untreated air leaks, tension pneumothorax, bronchopleural fistula, active hemoptysis, pulmonary haemorrhage, Large pulmonary bullae, intrathoracic obstruction from tumor or foreign body
* Unhealed dental, head, neck, ear, nose & throat, thoracic or upper gastro-intestinal tract surgery or trauma
* Unhealed broken ribs
* Esophageal varices
* Anxiety, Depression, history of Mental illness
* Dependence on positive pressure ventilation (i.e. 24/7 non-invasive ventilation).
* Cannot perform spirometry
* Enrollment in another interventional study
* Any medical condition for which the investigator deems the subject unable to participate in the study

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Constant Work Rate (CWR) Cardiopulmonary Exercise Test on cycle ergometer | at day 29
  Change from baseline in duration of constant work rate exercise testing (TLIM)

SECONDARY OUTCOMES:
Pulmonary functions test- FEV1 | at day 29 and 43
  Change from baseline in Forced Expiratory Volume in 1 Second (FEV1)
Pulmonary functions test- FRC | at day 29 and 43
  Change from baseline in Functional Residual Capacity (FRC)
Pulmonary functions test - FEF25-75 | at day 29 and 43
  Change from baseline in Forced Expiratory Flow Between 25% and 75% of Forced Vital Capacity (FEF25-75)
Pulmonary functions test- FVC | at day 29 and 43
  Change from baseline in Forced Vital Capacity (FVC)
COPD Assessment Test (CAT) | at day 29 and 43
  Change from baseline in score on CAT
Patients compliance rate to treatment | at day 29 and 43
  Compliance rate and treatment timings self-reported through subject diaries
CWR Cardiopulmonary Exercise Test on cycle ergometer- TLIM | at day 43
  Change from baseline in duration of constant work rate exercise testing (TLIM)
CWR Cardiopulmonary Exercise Test on cycle ergometer- VE | at day 29 and 43
  Changes from baseline in Expired Ventilation (VE)
CWR Cardiopulmonary Exercise Test on cycle ergometer- HR | at day 29 and 43
  Changes from baseline in Hart Rate (HR)
CWR Cardiopulmonary Exercise Test on cycle ergometer- SpO2 | at day 29 and 43
  Changes from baseline in Peripheral capillary oxygen saturation (SpO2)
CWR Cardiopulmonary Exercise Test on cycle ergometer- VT | at day 29 and 43
  Changes from baseline in Tidal Volume (VT)
CWR Cardiopulmonary Exercise Test on cycle ergometer- RR | at day 29 and 43
  Changes from baseline in Respiration Rate (RR)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Yarmolovsky, MD, Principal Investigator — Kaplan Medical Center, Israel